CLINICAL TRIAL: NCT00414778
Title: A Single-center, Open-label, Single and Multiple Oral Dose Study to Assess Safety and Pharmacokinetics of LHT344 in Chinese Healthy Subjects
Brief Title: Safety and Pharmacokinetics of LHT344 in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLHT344A2101
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: Healthy
Keywords: Safety, pharmacokinetics, oral, single dose, multiple dose, LHT344, Chinese, healthy subjects

INTERVENTIONS:
Drug: LHT344

SUMMARY:
The purpose of this study is to evaluate safety and pharmacokinetics of a single and multiple dose of LHT344 in 12 Chinese healthy subjects.

This study is not recruiting subjects in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking, male or female subjects age 18 to 45 years of age
* In good health as confirmed by past medical history, physical examination, electrocardiogram, laboratory tests and urinalysis on the screening and baseline evaluation
* Body mass index within the range of 19 to 24 kg/m2 and weigh at least 50 kg

Exclusion Criteria:

* Smokers
* Use of any prescription drugs within 4 weeks prior dosing, or over-the-counter medication (vitamins, herbal supplements, dietary supplements) within 2 weeks prior to dosing. Paracetamol is acceptable.
* Participation in any clinical investigation within 3 months prior to dosing.
* Donation or loss of 400 mL or more of blood within 12 weeks prior to first dosing required by local regulation.
* Significant illness within 2 weeks prior to dosing.
* A past personal or close family medical history of clinically significant cardiac abnormalities such as a myocardial infarction, angina, arterial fibrillation, arrhythmia or hypertension.
* History of
* fainting, low blood pressure upon standing, irregular heart beats
* acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated).
* clinically significant drug allergy, history or presence of atopic allergy (asthma, urticaria, eczematous dermatitis)
* known hypersensitivity to the study drug or similar drugs
* surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or may jeopardize the subject participation in the study
* immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.
* positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
* drug or alcohol abuse within the 12 months prior to study participation

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-10; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of single and repeat daily oral dose of LHT344 in Chinese healthy subjects

SECONDARY OUTCOMES:
Safety of single and repeat daily oral dose of LHT344 in Chinese healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, Beijing, China